CLINICAL TRIAL: NCT06241131
Title: Study on the Quality of Recovery From General Anesthesia With Desflurane for Fundus Surgery-A Single Center, Prospective, Randomized, Double-blind, Controlled Clinical Trial
Brief Title: The Quality of Recovery From General Anesthesia With Desflurane for Fundus Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ting Xu, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023-501
Record Dates: First submitted 2023-12-29; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Desflurane Anesthesia; Postoperative Recovery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- desflurane with remifentanil anesthesia (Experimental): Subjects were randomly assigned to the experimental group。In this group, desflurane was inhaled at a starting concentration of 1 MAC (Minimal Alveolar Concentration), and remifentanil 0.1 μg/kg/min was continuously pumped intravenously.
  Interventions: Drug: Desflurane Inhalant Product
- sevoflurane with remifentanil anesthesia (Active Comparator): Subjects were randomly assigned to the active comparator group。In this group, sevoflurane was inhaled at a starting concentration of 1 MAC, and remifentanil 0.1 μg/kg/min was continuously pumped intravenously.
  Interventions: Drug: Desflurane Inhalant Product

INTERVENTIONS:
Drug: Desflurane Inhalant Product — The Desflurane was inhaled at a starting concentration of 1 MAC, and remifentanil 0.1 μg/kg/min was continuously pumped intravenously.

SUMMARY:
The goal of this clinical trials to study and compare the effects of "desflurane with remifentanil anesthesia (study group)" and "sevoflurane with remifentanil anesthesia (control group)" for elective fundus surgery anesthesia. The main question it aims to answer are the characteristics of desflurane anesthesia in patients undergoing fundus surgery and to provide universal guidance for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II, patients aged 18-65 years old;
2. Fundus surgery to be performed under general anesthesia ;
3. The expected duration of surgery is about 30-120 min ;
4. BMI: 18-30 kg/m2 ;
5. Those who signed the informed consent form and volunteered to participate in this trial

Exclusion Criteria:

1. Patients with known or suspected genetic susceptibility to malignant hyperthermia;
2. Patients with history of asthma;
3. Patients with severe heart diseases (NYHA ≥ III, severe arrhythmia, etc.) and cerebral or pulmonary diseases, liver or kidney dysfunction; or with unstable vital signs;
4. Patients with history of long-term narcotic analgesics application, including sedative and antidepressant drugs;
5. Patients with history of psychotropic drug abuse within 3 months;
6. Patients with long-term alcohol abuse;
7. People with mental disorder and unable to communicate normally;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Recovery time | up to 1 hour
  The length of time from stopping anesthesia to patient recovery (opening eyes)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Xu, MD, Study Chair — Sichuan Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No